CLINICAL TRIAL: NCT00956436
Title: A Phase 1b, Open-Label Study of Sorafenib With BIIB022 in Subjects With Advanced Hepatocellular Carcinoma
Brief Title: Sorafenib With BIIB022 in Hepatocellular Carcinoma (HCC)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Terri Senta-McMillian, PRA, Int'l
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 212HC201
Record Dates: First submitted 2009-08-05; First posted 2009-08-11 (Estimated); Last update posted 2013-09-16 (Estimated); Status verified 2011-11

CONDITIONS: Hepatocellular Carcinoma
Keywords: Liver Cancer; Hepatocellular Carcinoma; Sorafenib; HCC; BIIB022; Open-Label; IGF-1R; Nexavar
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms; Insulin-Like Growth Factor I, Resistance To | interventions — BIIB022; Receptor Protein-Tyrosine Kinases; Antibodies, Monoclonal; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sorafenib Monotherapy (Experimental): Sorafenib Monotherapy
  Interventions: Drug: Sorafenib
- Sorafenib with BIIB022 (Experimental): Sorafenib with BIIB022
  Interventions: Drug: BIIB022

INTERVENTIONS:
Drug: BIIB022 — IV Q3W
  Other Names: IGF-1R; Liver Cancer; Hepatocellular Carcinoma; Monoclonal Antibody; Sorafenib; HCC; Nexavar
  Arms: Sorafenib with BIIB022
Drug: Sorafenib — Standard dosing of Sorafenib
  Other Names: HCC; Monoclonal Antibody; Hepatocellular Carcinoma; Liver Cancer; BIIB022; IGF-1R; Nexavar
  Arms: Sorafenib Monotherapy

SUMMARY:
This is a phase 1b, open-Label study of sorafenib with BIIB022 in subjects with advanced hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Histologically-confirmed advanced HCC with at least 1 target lesion measurable by modified RECIST.
* Child-Pugh score A5 or A6.
* ECOG Performance Status of ≤2.

Exclusion Criteria:

* Known central nervous system or brain metastases.
* Prior anti-IGF-1R therapy.
* Prior systemic therapy for advanced HCC. Prior local therapies are only permitted if subjects have documented disease progression according to modified RECIST.
* Concurrent anticancer therapy.
* History of myocardial infarction within 12 months prior to Day 1 or chronic heart failure.
* Acute hepatitis
* Fibrolamellar HCC

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-08; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of BIIB022 given once every 3 weeks in combination with sorafenib in subjects with advanced HCC. | 6 months

SECONDARY OUTCOMES:
To evaluate the PK profile of BIIB022 and sorafenib in this study population | 6 months
To assess the anti-tumor response in this study population | 6 months

CONTACTS AND LOCATIONS:
Locations (11):
- United States (6):
  - Resesarch Site, Denver, Colorado
  - Resesarch Site, Ocoee, Florida
  - Resesarch Site, Indianapolis, Indiana
  - Resesarch Site, Boston, Massachusetts
  - Resesarch Site, New York, New York
  - Resesarch Site, Norfolk, Virginia
- Resesarch Site, Singapore, Singapore
- Taiwan (3):
  - Resesarch Site, Tainan
  - Resesarch Site, Taipei
  - Resesarch Site, Taoyuan District
- Resesarch Site, Edgbaston, Birmingham, United Kingdom